CLINICAL TRIAL: NCT05975203
Title: Continuous Delivery Room Skin-to-skin-study for Moderate and Late Preterm Infants
Acronym: COSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Katrin Mehler, Associate Professor, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-1419
Record Dates: First submitted 2023-07-13; First posted 2023-08-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Preterm Birth; Mother-Infant Interaction; Infant Development
Keywords: preterm behavioral epigenetics; skin-to-skin contact
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention blinding of participant and care provider is not possible. The investigators are part of the care providing team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): After delivery the infant will be separated from the mother and placed on a primary care unit in another room to monitor the cardiopulmonary adaption for at least 20 minutes.
- skin-to-skin contact (Experimental): After delivery the infant will be put skin-to-skin on the mother's breast in comfort position for 60 minutes. The cardiopulmonary adaption will be monitored and supervised by the attending neonatologist and nurse.
  Interventions: Procedure: skin-to-skin contact

INTERVENTIONS:
Procedure: skin-to-skin contact — Immediately after delivery the infant will receive skin-to-skin contact with the mother.
  Arms: skin-to-skin contact

SUMMARY:
The goal of this randomized controlled trial is to compare the effect of direct skin-to-skin contact in moderate and late preterm infants. The main questions it aims to answer are:

* does skin-to-skin contact in moderate and late preterm infants influence gene expression in the stress signaling pathway?
* does skin-to-skin contact in moderate and late preterm infants improve the short- and long-term outcome?

Participants will either get immediate separation after vaginal birth or receive immediate skin-to-skin contact. Researchers will compare these two groups to answer the proposed questions.

DETAILED DESCRIPTION:
The planned study investigates prospectively the effect of early intervention (skin-to-skin contact in the delivery room) in moderate and late preterm infants on neonatal programming by determining gene expression in the stress signaling pathway. The working hypothesis of our project is that the intervention will affect gene expression in a way that subsequently leads to better long-term psycho-social and neurological development of these preterm infants. The study aims to improve the understanding of the correlation of behavioral and epigenetic parameters and prove the underlying hypothesis of a novel mechanistic link between immediate skin-to-skin contact in the delivery room and life-long stress tolerance.

ELIGIBILITY:
Inclusion Criteria:

* preterm birth between gestational age of 32 0/7 and 36 6/7 weeks
* vaginal delivery
* singleton
* informed consent before birth

Exclusion Criteria:

* malformations or syndromes of the infant
* resuscitation of the infant
* maternal psychological or severe physical illness
* lack of German language skills

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
gene expression in candidate genes of the stress signalling pathway | 36 to 72 hours after birth
  DNA will be extracted from peripheral white blood cells and mucosal epithelial cells. The expression of candidate genes of the stress signaling pathways are investigated. The candidate genes are glucocorticoid receptor (NR3C1), corticotropin releasing hormone (CRH), corticotropin-releasing hormone receptor 1 and 2 (CRHR1/2), serotonin transporter (slc6a4), vasopressin and brain-derived neurotrophic factor.
gene expression in candidate genes of the stress signalling pathway | corrected 6 months of age
  DNA and RNA will be extracted from mucosal epithelial cells. The expression of candidate genes of the stress signaling pathways are investigated. The candidate genes are glucocorticoid receptor (NR3C1), corticotropin releasing hormone (CRH), corticotropin-releasing hormone receptor 1 and 2 (CRHR1/2), serotonin transporter (slc6a4), vasopressin and brain-derived neurotrophic factor. Furthermore a whole-genome methylation will be analysed.
gene expression in candidate genes of the stress signalling pathway | corrected 24 months of age
  DNA will be extracted from mucosal epithelial cells. The expression of candidate genes of the stress signaling pathways are investigated. The candidate genes are glucocorticoid receptor (NR3C1), corticotropin releasing hormone (CRH), corticotropin-releasing hormone receptor 1 and 2 (CRHR1/2), serotonin transporter (slc6a4), vasopressin and brain-derived neurotrophic factor.

SECONDARY OUTCOMES:
mother-child-interaction | corrected 6 months of age
  Mother-child-interaction is investigated using Mannheim Rating Scales. Therefore a five-minute-videotape of the mother changing the infant's diapers and playing with the infant is used.
  Mannheim Rating Scales is a good validated standardized observation instrument. Stimulation and response from the mother as well from the infant are being recorded. Different communication channels can be used by mother and child (vocal, facial or motor).
  All behaviors are analysed at intervals of five seconds (event coding). Then the values are formed from the sum of the coded events.
  The scale ranges from 0 to 60. If there is no interaction, the scale is 0. If there is an interaction in each interval (every 5 seconds in a 5 minute videotape), the scale is 60. The mother-child interaction is better if the scale is higher.
General Movements | corrected 3 months of age
  The early infant development will be analyzed by general movements assessment by Prechtl. It is a validated diagnostic tool for the functional assessment of the young nervous system.
maternal depression | at inpatient discharge (assessed from 3 to 60 days of life), corrected 6 and 24 months of age
  Maternal depression is assessed with the German long form of the Center for Epidemiological Studies Depression Scale (CES-D). It is a self-report questionnaire to measure depressive symptoms and it consists of 20 questions. For each question the response choice are assigned point values (how often a symptom occurred during the last week). The point values are summed to a total measure score. The score ranges from 0 to 60. Zero points represents no symptoms of depression, a score of 15 or higher is interpreted to indicate a risk of depression.
social support | at inpatient discharge (assessed from 3 to 60 days of life), corrected 24 months of age
  Social support is assessed with the short version of the German questionnaire for social support (Fragebogen zur sozialen Unterstützung, questionnaire on social support) scale (F-SozU K-22).
  The questionnaire records the subjectively perceived or anticipated support from the social environment. There are 22 items and the test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). The scale ranges from a minimum of 22 points to a maximum of 110 points. The higher the score, the better the subjectively perceived or anticipated support.
socio-economic status | at inpatient discharge (assessed from 3 to 60 days of life)
  There will be a question to the household income per month and the parents' highest school-leaving certificate as well as the housing situation.
breastfeeding | at inpatient discharge (assessed from 3 to 60 days of life) and corrected six months of age
  There will be a question about breastfeeding.
impact of event scale | corrected 6 months of age
  Symptoms for post-traumatic stress is assessed with the impact of event scale - revised (IES-R). It is a self-report questionnaire and consists of 22 questions. For each question the response choice are assigned point values (how often a symptom occurred during the last week). The sub-scale values are summed by the corresponding sub-scale items. The three sub-scales are: intrusion, avoidance and hyperarousal. The overall result is calculated by a formula. The score ranges from -4,36 to 2,99. A result above 0 is interpreted to indicate a risk of post-traumatic stress disorder.
Parental Bonding | corrected 6 and 24 months of age
  Parental Bonding is assessed with the parental bonding questionnaire (PBQ). It consists of 25 items and each item is rated on a scale from 0 to 3 points (response range from "very like" to "very unlike"). There are four sub-scales and the point values of each sub-scale are summed to a total measure score. The four sub-scales are: impaired bonding, rejection and anger, anxiety about care, risk of abuse. The higher the score, the higher the risk of a disorder in each area of the sub-scale.
Parental Stress | corrected 6 and 24 months of age
  Parental stress is assessed with the German form of the parenting stress index (PSI).
  It consists of 48 items. The test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). There are 12 subscales, each consisting of 4 items and the points on the Likert scale are added. In each subscale there can be a minimum of 4 and a maximum of 20 points. The higher the score, the higher the parental stress.
reactivity of hypothalamic-pituitary-adrenal-axis | 36 to 72 hours after birth and corrected 24 months of age
  Salivary cortisol is measured before and 20 minutes after heel lance, respectively after a stressful testing. The saliva is collected by a small cotton roll, which is placed in the infants' mouth. The cortisol is assayed in duplicate using an immunoassay, which is a validated test.

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Mehler, PD Dr., Principal Investigator — University of Cologne
Locations (1):
- University hospital of Cologne, Department of Neonatology, Cologne, Northrhine-westfalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehler K, Hucklenbruch-Rother E, Trautmann-Villalba P, Becker I, Roth B, Kribs A. Delivery room skin-to-skin contact for preterm infants-A randomized clinical trial. Acta Paediatr. 2020 Mar;109(3):518-526. doi: 10.1111/apa.14975. Epub 2019 Sep 16. PMID 31423649
- [Background] Hucklenbruch-Rother E, Vohlen C, Mehdiani N, Keller T, Roth B, Kribs A, Mehler K. Delivery room skin-to-skin contact in preterm infants affects long-term expression of stress response genes. Psychoneuroendocrinology. 2020 Dec;122:104883. doi: 10.1016/j.psyneuen.2020.104883. Epub 2020 Sep 24. PMID 33027708